CLINICAL TRIAL: NCT02999672
Title: Phase II, Exploratory, Multicenter, Non Randomized, Single Agent Cohort Study to Determine Best Tumor Response With Trastuzumab Emtansine in HER2 Overexpressing Solid Tumors
Brief Title: A Study to Determine Best Tumor Response With Trastuzumab Emtansine in Human Epidermal Growth Factor Receptor 2 (HER2) Overexpressing Solid Tumors
Acronym: KAMELEON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO29694; 2015-001377-40 (EudraCT Number)
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Bladder Cancer; Pancreas Cancer; Cholangiocellular Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Pancreatic Neoplasms; Cholangiocarcinoma | interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (UBC) (Experimental): First six participants with locally advanced (unresectable and not treatable with curative intent) or metastatic UBC will initially receive Regimen A (trastuzumab emtansine at a dose of 2.4 mg/kg qw). An iDMC will assess the safety among the first six participants and decide whether dose will be switched to Regimen B (trastuzumab emtansine at a dose of 3.6 mg/kg q3w).
  Interventions: Drug: Trastuzumab Emtansine
- Cohort 2 (Pancreatic cancer/cholangiocarcinoma) (Experimental): First six participants with metastatic pancreatic cancer/cholangiocarcinoma will receive Regimen A (trastuzumab emtansine at a dose of 2.4 mg/kg qw). An iDMC will assess the safety among the first six participants and decide whether dose will be switched to Regimen B (trastuzumab emtansine at a dose of 3.6 mg/kg q3w).
  Interventions: Drug: Trastuzumab Emtansine

INTERVENTIONS:
Drug: Trastuzumab Emtansine — Trastuzumab emtansine will be administered as Regimen A (2.4 mg/kg qw via IV infusion) or Regimen B (3.6 mg/kg q3w via IV infusion) until unacceptable toxicity, withdrawal of consent, disease progression, or death, whichever occurs first.
  Other Names: Kadcyla

SUMMARY:
This multicenter, non-randomized, Phase II study will assess the efficacy, safety, and pharmacokinetics of trastuzumab emtansine in participants with HER2 overexpressing locally advanced (unresectable and not treatable with curative intent) or metastatic urothelial bladder cancer (UBC), locally advanced (unresectable and not treatable with curative intent) or metastatic pancreatic cancer/cholangiocarcinoma with advanced disease where cure is no longer possible and where no other treatment options are available anymore. Participants will receive intravenous (IV) infusion of trastuzumab emtansine as Regimen A (2.4 milligrams per kilogram [mg/kg], weekly [qw]) or Regimen B (3.6 mg/kg, every 3 weeks [q3w]) until unacceptable toxicity, withdrawal of consent, disease progression (PD), or death, whichever occurs first. Based on tolerability and safety aspects, steering committee and Independent Data Monitoring Committee (iDMC) will decide on expansion of the study to include more participants with other carcinoma types.

ELIGIBILITY:
Inclusion Criteria:

* Histologically centrally confirmed HER2-positive (immunohistochemistry [IHC]3+ in greater than or equal to [>/=] 30 percent [%] of tumor cells): locally advanced (unresectable and not treatable with curative intent), or metastatic UBC or locally advanced (unresectable and not treatable with curative intent) or metastatic pancreatic cancer/cholangiocarcinoma
* There must be no standard treatment options available for participants with the above HER2 overexpressing tumors and they must have undergone at least one prior platinum-based treatment for locally advanced (unresectable and not treatable with curative intent) or metastatic tumor (Note: for pancreatic cancer/cholangiocarcinoma, prior treatments are not required to be platinum-based.)
* Participant's lesion should be measurable according to RECIST V1.1 on diagnostic computed tomography (CT) scan/magnetic resonance imaging (MRI); Target lesion(s) should not have been previously irradiated
* At least one formalin-fixed paraffin-embedded (FFPE) biopsy of the primary tumor and/or from a metastatic site is required
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2
* No significant cardiac history and a current left ventricular ejection fraction (LVEF) >/=50%
* Adequate organ function
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Participants with previous exposure to HER2-targeted therapies in any setting
* Participants showing histologically confirmed focal HER2-expression, that is, less than (<) 30% of positively stained tumor cells
* Participants with brain metastasis as the sole site of metastatic disease and/or are symptomatic or require therapy to control symptoms
* Current uncontrolled hypertension (systolic greater than [>] 150 millimeters of mercury [mmHg] and/or diastolic >100 mmHg)
* Current unstable angina pectoris
* History of symptomatic congestive heart failure (CHF) of any New York Heart Association (NYHA) criteria or ventricular arrhythmia that requires treatment
* History of myocardial infarction within the last 6 months
* Peripheral neuropathy, Grade >/=3
* Current dyspnea at rest due to complications of advanced malignancy, or other diseases that require continuous oxygen therapy
* Current severe, uncontrolled systemic disease
* History of other malignancy within the last 5 years
* Concurrent, serious, uncontrolled infections or current known infection with human immunodeficiency virus (HIV), active hepatitis B and/or hepatitis C
* Known prior severe hypersensitivity to trastuzumab and trastuzumab emtansine or the excipients of the investigational medicinal product (IMP)
* Clinically significant bleeding within 30 days before enrollment
* Major surgical procedure or significant traumatic injury within 28 days prior to randomization or anticipation of the need for major surgery during the course of study treatment
* Concurrent participation in any other therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- Italy (5):
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - Irccs Ospedale San Raffaele;Oncologia Medica, Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO); Cure Mediche, Milan, Lombardy
  - IRCCS Istituto Oncologico Veneto (IOV); Oncologia Medica Prima, Padua, Veneto
  - A.O.U.I. VERONA-OSPEDALE POLICLINICO G.B. ROSSI BORGO ROMA;ONCOLOGIA MEDICA-d.U., Verona, Veneto
- Netherlands (4):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Amsterdam UMC Location VUMC, Amsterdam
  - UMCG, NL -groningen
  - Erasmus MC - Centrum, NL -rotterdam
- Narodny onkologicky ustav, Bratislava, Slovakia
- Spain (6):
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Duran i Reynals; Oncologia, Barcelona
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Regional Universitario Carlos Haya; Servicio de Oncologia, Málaga

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (UBC): First six participants with locally advanced (unresectable and not treatable with curative intent) or metastatic UBC initially received Regimen A (trastuzumab emtansine at a dose of 2.4 mg/kg qw). An iDMC assessed the safety among the first six participants and decided whether dose would be switched to Regimen B (trastuzumab emtansine at a dose of 3.6 mg/kg q3w).
- Cohort 2 (Pancreatic Cancer/Cholangiocarcinoma): First six participants with metastatic pancreatic cancer/cholangiocarcinoma received Regimen A (trastuzumab emtansine at a dose of 2.4 mg/kg qw). An iDMC assessed the safety among the first six participants and decided whether dose would be switched to Regimen B (trastuzumab emtansine at a dose of 3.6 mg/kg q3w).
Period: Overall Study
Arm/Group | Cohort 1 (UBC) | Cohort 2 (Pancreatic Cancer/Cholangiocarcinoma)
Started | 13 | 7
Completed | 0 | 0
Not Completed | 13 | 7
Not completed — Death | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 1
Not completed — Progressive Disease | 9 | 5
Not completed — Adverse Event | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (UBC) | Cohort 2 (Pancreatic Cancer/Cholangiocarcinoma) | Total
Number analyzed (Participants) | 13 | 7 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.4 (14.1) | 62.9 (7.2) | 59.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 12 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 9 | 7 | 16
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 7 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response (BOR) Assessed by the Investigator Using Response Evaluation Criteria in Solid Tumors [RECIST] 1.1).
Description: BOR was defined as having best objective response as complete response (CR) or partial response (PR), as assessed by investigator and confirmed at least 28 days after initial response, according to the Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1). CR was defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must decrease to normal (short axis less than [<] 10 millimeter [mm]). PR was defined as a 30% decrease in the sum of the diameters of the target lesions taking as a reference the baseline sum diameter. Percentage of participants with best overall response of CR or PR are reported.
Time Frame: Baseline up to PD/recurrence or death, whichever occurs first (up to approximately 18 months)
Population: Urothelial bladder cancer (UBC) and Pancreatic Cancer/Cholangiocarcinoma cohorts
Measure: Number; unit: Percentage of Treated Participants
Arm/Group | Cohort 1 (UBC) | Cohort 2 (Pancreatic Cancer/Cholangiocarcinoma)
Number analyzed (Participants) | 13 | 7
Percentage of Treated Participants
  CR | 0 | 0
  PR | 38.5 | 14.3

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was the time from inclusion in the study to the date of first documented PD or death from any cause, whichever occurred first. Participants without event were censored at the date of the last tumor assessment where non-progression was documented. If a participant received a second anti-cancer therapy without prior documentation of disease progression, the participant was censored at the date of last tumor assessment before starting new chemotherapy. PD was defined as at least a 20% increase in the sum of longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: Baseline up to PD/recurrence or death, whichever occurs first (up to approximately 18 months)
Population: Urothelial bladder cancer (UBC) and Pancreatic Cancer/Cholangiocarcinoma cohorts
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (UBC) | Cohort 2 (Pancreatic Cancer/Cholangiocarcinoma)
Number analyzed (Participants) | 13 | 7
Months | 2.20 [1.18 to 4.30] | 2.58 [1.31 to 9.99]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was determined as the time from beginning of treatment to death from any cause.
Time Frame: Baseline up to PD/recurrence or death, whichever occurs first (up to approximately 18 months)
Population: Urothelial bladder cancer (UBC) and Pancreatic Cancer/Cholangiocarcinoma cohorts
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (UBC) | Cohort 2 (Pancreatic Cancer/Cholangiocarcinoma)
Number analyzed (Participants) | 13 | 7
Months | 7.03 [3.75 to NA] — NA = NE= Not estimable. Upper limit of the 95 percent (%) confidence interval (CI) could not be calculated, as the study was terminated before a sufficient amount of data could be collected for accurate calculation. | NA [1.45 to NA] — NA = NE= Not estimable. Median and upper limit of the 95 percent (%) confidence interval (CI) could not be calculated, as the study was terminated before a sufficient amount of data could be collected for accurate calculation.

4. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious AEs (SAEs)
Description: Incidence, type and severity of all adverse events (AEs) and serious adverse events (SAEs), based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v4.03).
Time Frame: Baseline up to approximately 18 months
Population: Urothelial bladder cancer (UBC) and Pancreatic Cancer/Cholangiocarcinoma cohorts
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1 (UBC) | Cohort 2 (Pancreatic Cancer/Cholangiocarcinoma)
Number analyzed (Participants) | 13 | 7
Percentage of Participants
  AEs | 84.6 | 100
  Grade 1 AE | 7.7 | 14.3
  Grade 2 AE | 23.1 | 57.1
  Grade 3 AE | 30.8 | 28.1
  Grade 4 AE | 0 | 0
  Grade 5 AE | 23.1 | 0
  AE greater than Grade 3 | 53.8 | 28.6
  AE related to Trastuzumab Emtansine (TE) | 84.6 | 85.7
  SAEs | 46.2 | 28.6
  SAE related to TE | 0 | 0
  AE with fatal outcome | 23.1 | 0
  AE leading to discontinuation of TE | 23.1 | 0
  AE leading to modification of TE | 61.5 | 57.1
  AE of special interest | 0 | 0
  SAE of special interest | 0 | 0

5. Secondary Outcome: Percentage of Participants With Drug-induced Liver Injury Meeting Hy's Law Criteria
Description: Participants from both cohorts (UBC and Pancreatic cancer/cholangiocarcinoma) were analyzed for drug-induced liver injury following Hy's Law. Hy's Law criteria for potential drug-induced liver injury includes an elevated ALT (alanine aminotransferase) or AST (aspartate aminotransferase) in combination with either elevated bilirubin or clinical jaundice.
Time Frame: Baseline up to approximately 18 months
Population: Urothelial bladder cancer (UBC) and Pancreatic Cancer/Cholangiocarcinoma cohorts
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1 (UBC) | Cohort 2 (Pancreatic Cancer/Cholangiocarcinoma)
Number analyzed (Participants) | 13 | 7
Percentage of Participants | 0 | 0

6. Secondary Outcome: Plasma/Serum Concentrations of Trastuzumab Emtansine
Description: Samples for evaluation of trastuzumab emtansine, DM1, and total trastuzumab were obtained from all participants from both cohorts at specified time points.
Time Frame: Regimen A: predose (0 minutes [min]) and 15-30 min postinfusion on Days (D) 1, 8, 15 of Cycle (C) 1 and D1C4; predose on D1C2. Regimen B: predose and 15-30 min postinfusion on D1C1 and D1C4; predose on D1C2. 1 Cycle=21 days
Population: Urothelial bladder cancer (UBC) and Pancreatic Cancer/Cholangiocarcinoma cohorts.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 (UBC) | Cohort 2 (Pancreatic Cancer/Cholangiocarcinoma)
Number analyzed (Participants) | 13 | 7
ng/mL
  Predose, D1C1: number analyzed (Participants) | 13 | 1
  Predose, D1C1 | NA (NA) — Mean and Standard Deviation was not calculated due to below detection level. | NA (NA) — Due to low number of participants, standard deviation can not be calculated.
  15-30 min post-infusion, D1C1: number analyzed (Participants) | 13 | 6
  15-30 min post-infusion, D1C1 | 57.9 (16.1) | 52.3 (16.5)
  Predose, D8C1: number analyzed (Participants) | 6 | 4
  Predose, D8C1 | 8.27 (2.59) | 5.82 (1.96)
  15-30 min post-infusion, D8C1: number analyzed (Participants) | 6 | 3
  15-30 min post-infusion, D8C1 | 57.4 (12.0) | 50.3 (8.87)
  Predose, D15C1: number analyzed (Participants) | 5 | 1
  Predose, D15C1 | 14.8 (3.78) | 9.96 (NA) — Due to low number of participants, standard deviation can not be calculated.
  15-30 min post-infusion, D15C8: number analyzed (Participants) | 5 | 1
  15-30 min post-infusion, D15C8 | 59.3 (8.75) | 49.2 (NA) — Due to low number of participants, standard deviation can not be calculated.
  Predose, D1C2: number analyzed (Participants) | 11 | 5
  Predose, D1C2 | 10.5 (9.38) | 2.02 (2.08)
  Predose, D1C4: number analyzed (Participants) | 4 | 3
  Predose, D1C4 | 12.5 (8.63) | 11.7 (8.99)
  15-30 min post-infusion, D1C4: number analyzed (Participants) | 4 | 3
  15-30 min post-infusion, D1C4 | 62.5 (13.6) | 65.7 (10.5)

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 18 months
Description: An Adverse Event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure.
Arm/Group | Cohort 1 (UBC) | Cohort 2 (Pancreatic Cancer/Cholangiocarcinoma)
All-Cause Mortality (participants affected / at risk) | 7/13 | 1/7
Serious Adverse Events (participants affected / at risk) | 6/13 | 2/7
Other Adverse Events (participants affected / at risk) | 11/13 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (UBC) (N=13) | Cohort 2 (Pancreatic Cancer/Cholangiocarcinoma) (N=7)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (4) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Device-related sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (UBC) (N=13) | Cohort 2 (Pancreatic Cancer/Cholangiocarcinoma) (N=7)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 4 (5) | 2 (5)
Influenza like Illness (General disorders) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (2)
Pyrexia (General disorders) | 5 (6) | 3 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (5)
Abdominal pain, upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 2 (3)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Meralgia paraesthetica (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (4) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (2)
Malaise (General disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 3 (5)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The results represent the data up to primary completion date (10 April 2018). However, due to the early termination, the study was unable to fully address its primary and secondary objectives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT02999672/Prot_SAP_000.pdf